CLINICAL TRIAL: NCT03296254
Title: Comparison of Two Brief Mindfulness Intervention for Stress, Anxiety and Burnout in Mental Health Professionals: a Randomized Controlled Trial
Brief Title: Comparison of Two Brief Mindfulness Intervention for Stress, Anxiety and Burnout in Mental Health Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Educación a Distancia (Other)
Collaborators: Universidad de Ciencias Médicas de La Habana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 48817036RRI
Record Dates: First submitted 2017-09-18; First posted 2017-09-28 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Mental Health Wellness 1
Keywords: mindfulness; meditation; stress; burn-out; personality; randomized controlled trial
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: It is a 2-sequence, 2-period, 2-treatment crossover design with sequences AB and BA
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Course A (Experimental): Body Mindfulness Exercised followed by Sitting Mindfulness Exercises. Written material and sound recordings will be offered as support elements.
  Interventions: Behavioral: Sitting Mindfulness Exercises.; Behavioral: Body Mindfulness Exercises
- Course B (Experimental): Sitting Mindfulness Exercises followed by Body Mindfulness Exercises. Written material and sound recordings will be offered as support elements.
  Interventions: Behavioral: Sitting Mindfulness Exercises.; Behavioral: Body Mindfulness Exercises

INTERVENTIONS:
Behavioral: Sitting Mindfulness Exercises. — 5 weekly sessions of 2,5 hours/session of Sitting Mindfulness Meditation
Behavioral: Body Mindfulness Exercises — 5 weekly sessions of 2,5 hours/session of Body Scan and Mindful Movements

SUMMARY:
The aim of this study is to examine the effectiveness of two mindfulness interventions for stress, anxiety and burnout in mental health professionals. Participants will receive the treatments in reverse order: a brief intervention based on body-centered exercises and another brief intervention based on sitting meditation. It is hypothesized that both interventions will decrease stress and anxiety levels and professional burnout, with mindfulness body-centered exercises being at least as effective as mindfulness meditations.

DETAILED DESCRIPTION:
The aim of this study is to examine the effectiveness of two mindfulness interventions for stress, anxiety and burnout in mental health professionals. It is a 2-sequence, 2-period, 2-treatment crossover design with sequences AB and BA. Treatment A consists of a block of five sessions of bodyfulness exercises, whereas experimental treatment B consists of a block of five sessions of sitting mindfulness meditation exercises. In the sixth session, the exercise blocks will be exchanged. Each group will be composed of half the sample, with a initial sample of 130. The principal hypothesis is that both interventions will decrease stress and anxiety levels and professional burnout, with body-centered exercises being at least as effective as mindfulness sitting meditations. Secondarily, the personality type will be analyzed as a moderating variable in those variables in which the interventions will be effective. Third, a qualitative study will be conducted in order to analyze the perceptions of change and experiences in Cuban mental health professionals who are beginner meditators. This study will allow to understand the differential effectiveness of bodyfulness and midfulness and what types of personality may benefit most from different types of meditation interventions. Also, it will hell to get a deeper understanding of mindfulness practice in a new cultural context (i.e., Cuba). A previous pilot study will be conduct to investigate the acceptability and effectiveness of a culturally-adapted mindfulness-based intervention in Cuba.

ELIGIBILITY:
Inclusion Criteria:

* To be a full time mental health professional
* To be 18 years or older
* To be able to attend weekly sessions

Exclusion Criteria:

* To suffer a pathology that discourages participation in the study.
* Previous training in mindfulness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Stress at 5 weeks | Baseline, Post- treatment 5 weeks from baseline
  Stress measured using Seppo Aro Symptomatic Stress Scale
Change from Baseline Burnout at 5 weeks | Baseline, Post- treatment 5 weeks from baseline
  Burnout measured using Moreno Short Questionnaire of Burnout.
Change from Baseline Stress at 10 weeks | Baseline, Post- treatment 10 weeks
  Stress measured using Seppo Aro Symptomatic Stress Scale
Change from Baseline Stress at three-months follow-up | Baseline, Three-months follow-up
  Stress measured using Seppo Aro Symptomatic Stress Scale
Change from Baseline Burnout at 10 weeks | Baseline, Post- treatment 10 weeks
  Burnout measured using Moreno Short Questionnaire of Burnout.
Change from Baseline Burnout at at three-months follow-up | Baseline, Three-months follow-up
  Burnout measured using Moreno Short Questionnaire of Burnout.
Change from Baseline State Anxiety at 5 weeks | Baseline, Post- treatment 5 weeks from baseline
  State anxiety measured using State Anxiety Inventary IDARE
Change from Baseline State Anxiety at 10 weeks | Baseline, Post- treatment 10 weeks
  State anxiety measured using State Anxiety Inventary IDARE
Change from Baseline State Anxiety at three-months follow-up | Baseline, Three-months follow-up
  State anxiety measured using State Anxiety Inventary IDARE

SECONDARY OUTCOMES:
Sociodemographic data | Baseline
  Gender, age, marital status, professional status, years of mental health work, workplace, previous experience in related techniques.
The sixteen personality factor questionnaire | Baseline
  Cattell's 16 personality factors. This test uses a public domain scales from the Internation Personality Item Pool to measure the same traits.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Santed Germán, PhD, Study Director — Universidad Nacional a Distancia (España); Justo R Fabelo Roche, PhD, Study Chair — Universidad de Ciencias Médicas de La Habana (Cuba)
Locations (1):
- Justo Reinalod Fabelo Roche, La Habana, Cuba

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author, [Miguel A. Santed], upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] de Vibe M, Solhaug I, Tyssen R, Friborg O, Rosenvinge JH, Sorlie T, Halland E, Bjorndal A. Does Personality Moderate the Effects of Mindfulness Training for Medical and Psychology Students? Mindfulness (N Y). 2015;6(2):281-289. doi: 10.1007/s12671-013-0258-y. PMID 25798208
- [Background] Goodman MJ, Schorling JB. A mindfulness course decreases burnout and improves well-being among healthcare providers. Int J Psychiatry Med. 2012;43(2):119-28. doi: 10.2190/PM.43.2.b. PMID 22849035
- [Background] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Background] Ireland MJ, Clough B, Gill K, Langan F, O'Connor A, Spencer L. A randomized controlled trial of mindfulness to reduce stress and burnout among intern medical practitioners. Med Teach. 2017 Apr;39(4):409-414. doi: 10.1080/0142159X.2017.1294749. Epub 2017 Feb 28. PMID 28379084
- [Background] Irving JA, Dobkin PL, Park J. Cultivating mindfulness in health care professionals: a review of empirical studies of mindfulness-based stress reduction (MBSR). Complement Ther Clin Pract. 2009 May;15(2):61-6. doi: 10.1016/j.ctcp.2009.01.002. Epub 2009 Feb 28. PMID 19341981
- [Background] Morse G, Salyers MP, Rollins AL, Monroe-DeVita M, Pfahler C. Burnout in mental health services: a review of the problem and its remediation. Adm Policy Ment Health. 2012 Sep;39(5):341-52. doi: 10.1007/s10488-011-0352-1. PMID 21533847
- [Derived] Ruiz-Iniguez R, Carralero Montero A, Burgos-Julian FA, Fabelo Roche JR, Santed MA. Comparison of two brief mindfulness interventions for anxiety, stress and burnout in mental health professionals: a randomised crossover trial. Front Psychol. 2023 May 12;14:1160714. doi: 10.3389/fpsyg.2023.1160714. eCollection 2023. PMID 37251062
- [Derived] Ruiz-Iniguez R, Carralero Montero A, Burgos-Julian FA, Fabelo Roche JR, Santed MA. Interactions between Personality and Types of Mindfulness Practice in Reducing Burnout in Mental Health Professionals. Int J Environ Res Public Health. 2021 Jun 22;18(13):6721. doi: 10.3390/ijerph18136721. PMID 34206446
- See also: Investigations at the National Distance Education University — http://portal.uned.es/portal/page?_pageid=93,25453043&_dad=portal&_schema=PORTAL